CLINICAL TRIAL: NCT06759220
Title: Hystrolaparosciopic Findings in Infertile Women with Secondary Infertility
Brief Title: Hystrolaparoscopic Findings in Infertile Women with Previous Uterine Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Ali Ramadan, Dalia Ali Ramadan, Assiut University
Other Study IDs: Laparoscopy in infertility
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-09

CONDITIONS: Hystrolaparoscopic Findings in Infertile Women with Previous Uterine Surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1. to determine the rate and pattern of abnormal laparoscopic finding among the infertile women with history of previous uterine surgery.
2. To detemine the rate and pattern of abnormal hysteroscopic finding among infertile women with with history of previous uterine sergery
3. to evaluate the value of doing combined laparoscopy and hysteroscopy in infertile women with with history of previous uterine surgery.
4. To determine possible risk factors of pelvic adhesions detected during laparoscopy.
5. To determine possible risk factors causing cs niche.

DETAILED DESCRIPTION:
nfertility(1), which refers to the inability of a couple to conceive after one year of regular unprotected sexual intercourse, is the commonest indication for gynacological consultation. primary infertility - where someone who's never conceived a child in the past. secondary infertility(2) - where someone has had 1 or more pregnancies in the past, but is having difficulty conceiving again.there are many causes for infertility. (3)uterine causes as uterine fibroids or malformations.tubal factors as tuboperitoneal adhesions,unilateral or bilateral proximal occlusion unilateral or bilateral hydrosalpinx or pyosalpinx.Ovarian factors ovarian cyst,polycystic ovaries.pelvic causes as adhesions ,endometriosis and miscellaneous. laparoscopy can be used as the gold standard diagnostic tool which allows direct visualization of all pelvic organs. It also helps in detailed assessment of fallopian tubes. The advantage behind using laparoscopy is that the treatment of certain conditions such as tubal obstruction, endometriosis, and pelvic adhesions can be done at the same time during diagnosis. If needed, laparoscopic chromopertubation can also be done for tubal patency during the same sitting. (4)Hysteroscopy is the direct visualization of the uterine cavity using an endoscope. Uterine cavity evaluation is very much needed to do achieve total infertility workup. Uterine abnormalities are present among 10-15% of couples who seek treatment of infertility. For evaluation of endometrial factors,(5) hysteroscopy considered to be a gold standard. Diagnostic h hysteroscopy can detect uterine anomalies which remain undetected in USG and other routine investigations.

Many studies reported the occurrence of pelvic adhesions following cesarean section with its related consequences.

pelvic adhesions may affect both reproductive system anatomy and function, causing various associated conditions. Pelvic adhesions may cause secondary infertility, which might be due to dyspareunia, disturbing tubo-ovarian relationship, or disturbing peristaltic movement of fallopian tube.

ELIGIBILITY:
Inclusion Criteria:

* All women between20 to 35 yrs old with secondary infertiliy for 2 years
* Women with previous uterine surgery

Exclusion Criteria:

* Female with major medical illness(Uncontrolled daibetes, cardiac diseases, uncontrolled thyroid disorders)
* Abnormal semen parameter of the husband.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females
Study Population: Infertile women between age of 20to 35yr with previous uterine surgeries
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-21 (Estimated); Primary Completion 2027-03-21 (Estimated); Study Completion 2028-09-21 (Estimated)

PRIMARY OUTCOMES:
Primary (main): rate and pattern of abnormal laparoscopic and hysteroscopic findings in infertile women with previous uterine surgery | Baseline
  Primary (main): rate and pattern of abnormal laparoscopic and hysteroscopic findings in infertile women with previous uterine surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Women's health hospital Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibekwe PC, Udensi AM, Imo AO. Hysterosalpingographic findings in patients with infertility in South eastern Nigeria. Niger J Med. 2010 Apr-Jun;19(2):165-7. doi: 10.4314/njm.v19i2.56510. PMID 20642082
- [Background] Bukar M, Mustapha Z, Takai UI, Tahir A. Hysterosalpingographic findings in infertile women: a seven year review. Niger J Clin Pract. 2011 Apr-Jun;14(2):168-70. doi: 10.4103/1119-3077.84008. PMID 21860133
- [Background] Bello TO. Tubal abnormalities on hysterosalpingography in primary and secondary infertility. West Afr J Med. 2006 Apr-Jun;25(2):130-3. doi: 10.4314/wajm.v25i2.28263. PMID 16918185
- [Background] Adesiyun AG, Ameh CA, Eka A. Hysterosalpingographic tubal abnormalities and HIV infection among black women with tubal infertility in sub-Saharan Africa. Gynecol Obstet Invest. 2008;66(2):119-22. doi: 10.1159/000128600. Epub 2008 Apr 29. PMID 18446041